CLINICAL TRIAL: NCT03061344
Title: Endoscopic Buccal Mucosal Graft Urethroplasty or Bladder Neck Reconstruction
Brief Title: Liquid Buccal Mucosa Graft Urethroplasty
Acronym: LBMG
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Dmitriy Nikolavsky, Assistant Professor, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUNYUpstateMU
Record Dates: First submitted 2016-08-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- liquid buccal mucosa graft (Experimental): DVIU treated with liquid buccal mucosal graft; endoscopic injection of morcellated buccal mucosal graft mixed with fibrin glue
  Interventions: Biological: DVIU treated with liquid buccal mucosal graft

INTERVENTIONS:
Biological: DVIU treated with liquid buccal mucosal graft — DVIU treated with liquid buccal mucosal graft; internal urethrotomy for urethral stricture followed by injection of morcellated buccal mucosal graft mixed with fibrin glue (Tisseel, Baxter)

SUMMARY:
Study Objectives The current definitive treatment options for urethral stricture disease include endoscopic urethrotomy known as Direct Vision Internal Urethrotomy (DVIU) or open reconstruction known as urethroplasty (1-6). The purpose of this study is to determine feasibility of endoscopic-only repair of urethral stricture or bladder neck contracture using a combination of existing surgical techniques of internal urethrotomy (or bladder neck incision) augmented by buccal mucosal graft.

DETAILED DESCRIPTION:
Background and Rationale There are two definitive treatment options for urethral strictures: DVIU and open urethroplasty. DVIU is an endoscopic procedure considered to be minimally invasive, but also with a high failure rate of 60-92%. The repeated DVIUs are reported to have even higher failure rates. On the other hand, open urethroplasty, considered a gold standard for reconstruction, is invasive, requires incision of the perineum or urethra, leaves a life-long scar, and has long term success rates of 74-95%. The details of DVIU and open urethroplasty are discussed below.

DVIU involves passing a cystoscope into the urethra to the level of stricture and incising the stricture longitudinally to create a wide passage to the level of normal urethra on the proximal side. The hope is to cut through the scar to the level of healthy underlying tissue and in the process of healing to populate the cut surface with healthy urethral epithelium (or at least to stabilize the scar in open configuration). In most cases, the scarring recurs faster than epithelization and most strictures recur after DVIU within 7-8 months. Studies show the strictures after traditional repeat DVIU are longer and require more involved reconstruction than strictures in patients without prior instrumentation.

Open urethroplasty for urethral strictures or bladder neck contractures usually involves longitudinal incision of the urethra (from outside in) and augmentation of the incised part with a strip of harvested Buccal Mucosal Graft (BMG). The goal of the operation is to create a wide urethral lumen for the patient to be able to pass urine without obstruction.

The first step of the procedure for DVIU and open reconstruction are nearly the same: a longitudinal incision of the scarred portion of the urethra. The difference is in the second part: covering the defect with buccal mucosal graft as in open urethroplasty vs leaving the incision uncovered and exposed to passage of urine.

Investigators of this study hereby propose to combine the minimally invasive technique of the DVIU with the technique of augmenting the incised stricture (or bladder neck contracture) using buccal mucosal graft placed endoscopically by means of application of liquid suspended graft. A similar, but more invasive technique was reported by Seith et al in 2012 performed in 12 patients with the exception of need for small open perineal incision for graft fixation. A purely endoscopic skin graft placement into urethra was reported by Naude in 1998 in 53 patients with 95% success rate at 2 years follow up. While he has not made actual incisions, his approach required percutaneous perineal needle placement for graft delivery and a specialized device for graft delivery and graft fixation. The procedure proposed for current trial is purely endoscopic with buccal graft placement and fixation augmented by fibrin glue. This type of fibrin glue sealant is readily available and widely used in General Surgery, Plastic Surgery and in Urology specifically for urethral reconstruction). This will allow for significantly less invasive procedure, shorter procedure time, absence of traditional perineal incision or needle puncture, and earlier return home (same day vs 1-3 days), earlier catheter removal (5-7 days vs 21 days) and earlier return to regular activities (1 week vs 6 weeks).

Overall, the aim is to improve the outcomes of traditional endoscopic procedure while eliminating morbidity of the open reconstruction with added benefits of earlier convalescence and health care savings from decreased surgical morbidity and shortened hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Male >18 years of age
* bulbar urethral stricture
* bladder neck contracture

Exclusion Criteria:

* <18 years old
* developmental delay
* incarcerated individuals,
* history of prior urethroplasty
* history of cerebrovascular diseases (prior stroke, MI)
* history of deep vein thrombosis
* history of pulmonary embolism
* history of clotting disorders
* factor 5 Leiden
* antiphospholipid antibody syndrome
* prothrombin gene mutation
* protein S deficiency
* protein C deficiency
* dysfibrinogenemia
* polycythemia vera
* essential thrombocytosis
* untreated malignancy
* hypercoagulable state

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Voiding Surgical Outcomes: Stricture Recurrence | 3 years
  The ultimate outcome of this procedure is number of patients successfully treated without need for re-intervention (such as need for urethral dilation, endoscopic manipulation or open reconstruction). Recurrence of stricture will be reported as number of events. To detect stricture recurrence, patients will be monitored with: peak urine flow (milliliters per second) and post-void residuals (milliliters) and will be assessed post- operatively at every visit up to three years Flexible cystoscopy will be offered to patients at one year follow up or at any time point if there is suspicion of stricture recurrence based on patients complaints (reported as number of recurrences).

SECONDARY OUTCOMES:
Immediate Perioperative Outcomes | Day of surgery
  This is a composite outcome measure consisting of the following measures: duration of surgery (time in minutes), immediate postoperative complications: bleeding requiring blood transfusion (units of transfused blood), cerebrovascular complications reported as number of events (stroke, myocardial infarctions, pulmonary emboli) , problems with anesthesia (inability to extubate, need to re-intubate reported as number of each events), allergic reactions including anaphylaxis (number) and, duration of hospital stay (days).
Short-term Postoperative Outcomes | Up to 90 days
  This is a composite outcome measure consisting of the following measures: Urinary Tract Infection (number of infections requiring treatment), Sepsis (number of events), unscheduled ER visits (number), readmissions for hospital stay (number of events).
Patient Satisfaction | Post-operative up to 3 years follow up
  Global Response Assessment questionnaire will be given to patients at every visit to assess overall satisfaction with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Nikolavsky, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No